CLINICAL TRIAL: NCT06813833
Title: Image Markers and Transcriptome Profiles: an Exploratory Study of Optical Coherence Tomography and Tape Strips for Basal Cell Carcinoma
Brief Title: Transcriptomic Analysis and Optical Coherence Tomography Combined for Patients With Basal Cell Carcinoma
Acronym: RNA-OCT-BCC
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Merete Haedersdal, Professor, Chief Physician, DMSc, PhD, Bispebjerg Hospital
Other Study IDs: H-24060543; H-24060543 (Other: The Regional Research Ethics Committees)
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Basal Cell Carcinomas
Keywords: Basal Cell Carcinoma; Optical Coherence Tomography; Transcriptomics; Tape strip; Skin Cancer; Keratinocyte Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tape strips for transcriptomic analysis of BCC and healthy skin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to learn if tape strip for transcriptomic (RNA) analysis and optical coherence tomography (OCT) combined can optimize noninvasive management of basal cell carcinoma (BCC) patients.

The main question of the study is to examine if the combination of these two techniques, transcriptomic and OCT, can improve noninvasive detection of human BCCs.

All included patients will undergo 1) an OCT scan and 2) a tape strip collection for transcriptomic analysis from the same BCC.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years with clinical suspicious BCC for inclusion in the study and BCC histopathology diagnosis for inclusion in our analysis.

Exclusion Criteria:

* Patients with a BCC in areas not amenable to OCT (e.g., around the eye).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histology verified basal cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Association between tape strip and OCT | Single time point at baseline examination
  The association between BCC-specific image marker profiles from OCT and BCC-specific transcriptomic profiles from tape strips, in histopathologically confirmed BCC patients.

CONTACTS AND LOCATIONS:
Overall Officials: Merete Haedersdal, Professor, MD, DMSc, PhD, Principal Investigator — Department of Dermatology, Copenhagen University Hospital - Bispebjerg, Copenhagen, Denmark
Locations (1):
- Department of Dermatology, Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided